CLINICAL TRIAL: NCT01457131
Title: Phase I/II Study of Metastatic Cancer That Expresses NY-ESO-1 Using Lymphodepleting Conditioning Followed by Infusion of Gene Engineered Lymphocytes Cotransduced With Genes Encoding IL-12 and Anti-NY ESO-1 TCR
Brief Title: Modified White Blood Cells That Secrete IL-2 and Express a Protein That Targets the ESO-1tumor Protein for Metastatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120006; 12-C-0006
Record Dates: First submitted 2011-10-12; First posted 2011-10-21 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2013-08-02

CONDITIONS: Metastatic Cancer; Metastatic Melanoma; Metastatic Renal Cancer
Keywords: Metastatic Cancer; Immunotherapy; Gene Therapy; Metastatic Melanoma; Metastatic Kidney Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Kidney Neoplasms | interventions — fludarabine; Cyclophosphamide; Interleukin-12; Adenosine Monophosphate

INTERVENTIONS:
Drug: Fludarabine — 50 mg/m2, IV(in the vein)on day 5 of each 25 day cycle
Drug: Cyclophosphamide — 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days
Other: IL-12 & Anti-NY ESO1 TCR PBL — 10(7) cells to 3 X 10(10) cells

SUMMARY:
Background:

- A new cancer treatment involves collecting white blood cells from an individual, modifying them to secrete IL-2 and target the ESO-1 protein expressed on some cancers, and returning them to the body. The cells may then be able to seek out the cancer cells and destroy them. Some kinds of cancer contain a protein called ESO-1, which is found on the surface of the cells. Doctors want to modify white blood cells to have an anti-ESO-1 effect, and use them to treat the cancer that has the ESO-1. In addition to adding genes that target the ESO-1 protein to the cells, the genes for IL-12 are added to the cells. IL-12 is a protein that stimulates the immune system. This type of therapy is called gene transfer.

Objectives:

- To test the safety and effectiveness of anti-ESO-1/IL-12 white blood cells against metastatic cancer.

Eligibility:

- Individuals at least 18 years of age who have metastatic cancer that expresses ESO-1 and has not responded to standard treatments.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood tests and imaging studies.
* Participants will have leukapheresis about a month before the treatment to collect white blood cells.
* They will have chemotherapy 5 days before the treatment to suppress the immune system, and prepare the body for the anti-ESO-1/IL-12 cells.
* The anti-ESO-1/IL-12 cells will be given as an infusion.
* Participants will be monitored in the hospital during their recovery from the treatment.
* Participants will have regular followup exams every 1 to 6 months. The exams will include blood tests, imaging studies, and other studies.

Due to toxicities seen with the regimen, it was decided not to pursue the phase 2 portion of the study.

DETAILED DESCRIPTION:
Background:

* In prior trials we have shown that adoptive transfer of lymphocytes, transduced with a T cell receptor (TCR) that recognizes the NY-ESO-1 antigen, can mediate regression of metastatic cancer, though responses are often transient, and complete responses are rare.
* Interleukin-12 (IL-12) is an important immunostimulatory cytokine. We have constructed a retroviral vector that contains an inducible single chain IL-12 driven by an NFAT responsive promoter which can be used to mediate transfer of this gene into anti-tumor lymphocytes. This construct enables the secretion of IL-12 following stimulation of the TCR.
* Transduction of the IL-12 gene into mouse anti-tumor lymphocytes results in a profound increase in the ability of these lymphocytes to mediate tumor regression following administration to tumor bearing mice. These cells have a profound advantage in inducing anti-tumor responses because very few cells are needed and there is no requirement for the concomitant administration of interleukin-2 (IL-2) as is the case for conventional cell transfer immunotherapies.
* Based on these studies we have now used a retrovirus that encodes an inducible human single chain IL-12 driven by an NFAT responsive promoter and a retrovirus that encodes an anti-NY-ESO-1 TCR to cotransduce autologous lymphocytes for the treatment of patients with metastatic cancer that expresses the NY-ESO-1 antigen.

Objectives:

Primary objectives:

* To evaluate the safety of the administration of IL-12 and anti-NY-ESO-1 engineered lymphocytes in patients receiving a non-myeloablative conditioning regimen.
* To determine if the administration of the transduced lymphocytes to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer.

Secondary objective:

- To determine the in vivo survival of cotransduced gene-engineered cells.

Eligibility:

Patients who are 18 years of age or older must have

* Metastatic cancer whose tumors express the ESO antigen;
* ECOG performance status 0 or 1;

Design:

* Autlogous lymphocytes will be cotransduced with retroviral vectors, encoding IL-12 and anti- NY-ESO-1 TCR.
* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of IL-12/anti-ESO TCR gene-transduced lymphocytes.
* Patients will undergo complete evaluation of tumor with physical examination, CT of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment. If the patient has SD or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will continue to be followed with this evaluation every 3-4 months until off study criteria are met.
* The study will be conducted using a Phase I/II optimal design. The protocol will proceed in a phase 1 dose escalation design. Initially, the protocol will enroll 1 patient in each of the first 3 dose cohorts unless that patient experiences a dose limiting toxicity (DLT). Following cohort 3, all subsequent cohorts will proceed in a phase 1 dose escalation design, with 5 cohorts of n=3. Should a single patient experience a DLT due to the cell transfer at a particular dose level, additional patients would be treated at that dose to confirm that no greater than 1/6 patients have a DLT prior to proceeding to the next higher level. If a level with 2 or more DLTs in 3-6 patients has been identified, three additional patients will be accrued at the next-lowest dose, for a total of 6, in order to further characterize the safety of the maximum tolerated dose (MTD) prior to starting the phase II portion. If a DLT occurs in the first cohort, that cohort will be expanded to 6 patients. If 2 DLTs are encountered in this cohort, the study will be terminated.
* Once the MTD has been determined, the study then will proceed to the phase II portion using a phase II optimal design where initially 21 evaluable patients will be enrolled in each of 2 cohorts. If 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled.
* The objective will be to determine if the combination of lymphocyte depleting chemotherapy, and IL-12/ESO TCR gene engineered lymphocytes is associated with a complete response rate that can rule out 5% (p0=0.05) in favor of a modest 20% PR + CR rate (p1=0.20).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic cancer that expresses ESO as assessed by one of the following methods: RT-PCR on tumor tissue, or by immunohistochemistry of resected tissue, or serum antibody reactive with ESO. Metastatic cancer diagnosis will be confirmed by the Laboratory of Pathology at the NCI.
  2. Patients with melanoma or renal cell cancer must have previously received high dose IL-2 and have been either non-responders (progressive disease) or have recurred. Patients with other histologies, must have previously received systemic standard care (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.
  3. Greater than or equal to 18 years of age.
  4. Willing to sign a durable power of attorney
  5. Able to understand and sign the Informed Consent Document
  6. Clinical performance status of ECOG 0 or 1.
  7. Life expectancy of greater than three months.
  8. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
  9. Patients must be HLA-A*0201 positive
  10. Serology:

      1. Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
      2. Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
  11. Hematology:

      1. Absolute neutrophil count greater than 1000/mm3 without the support of filgrastim.
      2. WBC (> 3000/mm(3)).
      3. Platelet count greater than 100,000/mm(3).
      4. Hemoglobin greater than 8.0 g/dl.
  12. Chemistry:

      1. Serum ALT/AST less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert s Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  13. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
  14. Six weeks must have elapsed since any prior anti-CTLA4 antibody therapy to allow antibody levels to decline.
  15. Patients who have previously received any anti-CTLA4 antibody and have documented GI toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Previous treatment with IL-12.
2. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
3. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
6. Concurrent systemic steroid therapy.
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. History of coronary revascularization or ischemic symptoms
9. Any patient known to have an LVEF less than or equal to 45%.
10. Documented LVEF of less than or equal to 45% tested in patients with:

    1. History of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
    2. Age greater than 60 years old
11. Documented FEV1 less than or equal to 60% predicted tested in patients with:

    1. A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
    2. Symptoms of respiratory dysfunction

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10-06; Primary Completion 2013-08-07 (Actual); Study Completion 2013-08-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the IL-12 and anti-NY-ESO-1 engineered PBL in patients receiving a non-myeloablative conditioning regimen, and to determine if patients with metastatic cancer will have clinical tumor regression following this regimen. | 4 years

SECONDARY OUTCOMES:
To determine the in vivo survival of cotransduced gene-engineered cells. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chen YT, Scanlan MJ, Sahin U, Tureci O, Gure AO, Tsang S, Williamson B, Stockert E, Pfreundschuh M, Old LJ. A testicular antigen aberrantly expressed in human cancers detected by autologous antibody screening. Proc Natl Acad Sci U S A. 1997 Mar 4;94(5):1914-8. doi: 10.1073/pnas.94.5.1914. PMID 9050879
- [Background] Dudley ME, Yang JC, Sherry R, Hughes MS, Royal R, Kammula U, Robbins PF, Huang J, Citrin DE, Leitman SF, Wunderlich J, Restifo NP, Thomasian A, Downey SG, Smith FO, Klapper J, Morton K, Laurencot C, White DE, Rosenberg SA. Adoptive cell therapy for patients with metastatic melanoma: evaluation of intensive myeloablative chemoradiation preparative regimens. J Clin Oncol. 2008 Nov 10;26(32):5233-9. doi: 10.1200/JCO.2008.16.5449. Epub 2008 Sep 22. PMID 18809613
- [Background] Lethe B, Lucas S, Michaux L, De Smet C, Godelaine D, Serrano A, De Plaen E, Boon T. LAGE-1, a new gene with tumor specificity. Int J Cancer. 1998 Jun 10;76(6):903-8. doi: 10.1002/(sici)1097-0215(19980610)76:63.0.co;2-1. PMID 9626360